CLINICAL TRIAL: NCT03020654
Title: The Use of Virtual Reality for the Treatment of Visual Vertigo.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH19451; 5375 (Other: University of Manchester)
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2017-10

CONDITIONS: Treatment of Visual Vertigo

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Virtual environment with fast moving objects these are graded in intensity from 1-7. Participants complete head and eye exercises within the environment using focus points such as benches and lanterns for a six week treatment program.
  Interventions: Other: Virtual environment with fast moving objects
- Control group (Active Comparator): Virtual environment with no movement graded at grade 0. Participants complete head and eye exercises within the environment using focus points such as benches and lanterns for a six week treatment program.
  Interventions: Other: Virtual environment with no movement

INTERVENTIONS:
Other: Virtual environment with fast moving objects — A beach/park environment with graded moving objects, the individual will complete head and eye exercises.
  Arms: Treatment group
Other: Virtual environment with no movement — A beach/park environment with static objects, the individual will complete head and eye exercises.
  Arms: Control group

SUMMARY:
This study investigates the use of virtual environments presented on a head mounted display for the rehabilitation of those suffering with visual vertigo.

The control group and treatment groups will be presented with two different sets of environments and be given the same head and eye exercises to complete within the environment. They will also be provided with at home exercises to complete.

DETAILED DESCRIPTION:
Visual vertigo occurs after the balance system suffers damage (e.g after a viral infection such as labyrinthitis). This causes an over-reliance on the eyes to maintain balance which causes disorientation in busy environments such as the supermarket. The treatment involves trying to desensitise the individual to visually stimulating situations. Further head and eye exercises are completed alongside the exposure to overcome the damage done to the balance system.

ELIGIBILITY:
Inclusion Criteria:

* Those who have been diagnosed with visual vertigo and have scored a significant level on the Situational Characteristic Questionnaire (over 0.74 as per Pavlou et al., 2006).

Exclusion Criteria:

* Those with or under investigation for epilepsy.
* Those who have been determined to have no or limited balance function in both ears.
* Those with reduced visual acuity that will leave them unable to view the 3D effects of the head mounted display.
* Those with severe mental health disorders e.g. psychosis, paranoid disorders, bipolar disorder or a history of substance abuse.
* Severe neck pain/ restricted movement.
* Previous treatment for visual vertigo.
* Those with an fluctuating vestibular disorder such as Ménière's disease or vestibular migraine.
* Those with untreated Benign Paroxymal Positional Vertigo (BPPV).
* Those with a significant brain injury, or head injury that results in a central vestibular disorder.
* Those with an arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change in scoring on the Situational Characteristic Questionnaire | Week 1 and Week 6
  A measure of visual vertigo symptom level

SECONDARY OUTCOMES:
Change in scoring on the PHQ-9 Questionnaire from week one to six | Week 1 and Week 6
  A measure of depression symptom level
Change in scoring on the GAD-7 Questionnaire from week one to six | Week 1 and Week 6
  A measure of anxiety symptom level

OTHER OUTCOMES:
Subjective questionnaire | Week 6
  A likert scale based questionnaire assessing acceptability of treatment
Change in head tracking observed at each weekly session for six weeks through numerical data extracted from the headset to show displacement of the head in the x, y and z planes of movement. | Week 1, 2, 3, 4, 5 and 6
  Analysis of the head movement within each environment each week to see if there is any improvement

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty M Walker, BSc, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No